CLINICAL TRIAL: NCT00145366
Title: Pretreatment With Recombinant Human Thyrotropin (rhTSH) for the Effect on Thyroid Size and Function, and for the Effect of Radioiodine Treatment in Patients With Nodular Goiter. Prospective, Randomized Double-blinded Trials.
Brief Title: rhTSH, Thyroid Size, and Radioiodine Therapy in Benign Goiter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2009-04

CONDITIONS: Benign Nontoxic and Toxic Goiter; Graves' Disease
Keywords: Benign nontoxic and toxic goiter; rhTSH; 131I; goiter reduction; 131I kinetic; thyroid size; patient satisfaction; adverse effects; BRT; Graves' disease
MeSH Terms: conditions — Graves Disease; Patient Satisfaction | interventions — Thyrotropin Alfa

INTERVENTIONS:
Drug: Recombinant human thyrotropin (Thyrogen)

SUMMARY:
The trials in this protocol deals with the effect of pretreatment with rhTSH on radioiodine treatment of thyroid size and function, in patients with nontoxic and toxic nodular goiter. It is an introduction of a novel principle, based on prospective, randomized double blind investigations. Attached to this, we investigate the acute effects of rhTSH on thyroid size (measured by ultrasonography), both in healthy individuals and in patients with nontoxic nodular goiter. Thus, the investigations are divided into 4 categories listed below:

1. Prospective randomized double blind study of pretreatment with 0.3 mg recombinant human TSH for the effect of radioiodine in nontoxic multinodular goiter.
2. Prospective randomized double blind study of the pretreatment with 0.3 mg recombinant human TSH for the effect of radioiodine on thyroid size and function in patients with a very large (>100 ml) nontoxic or toxic goiter.
3. Does administration of 0.9 mg recombinant human TSH affect thyroid function and volume in healthy individuals? A randomized double-blind cross-over trial.
4. Does administration of 0.3 mg recombinant human TSH affect thyroid function and volume in healthy individuals and in patients with multinodular non-toxic goiter? A randomized double-blind cross-over trial.

   As a final note we investigate, in a pilot-study;
5. The influence of rhTSH on thyroid radioiodine uptake in patients with hyperthyroidism treated with continuous block-replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with an intact thyroid gland
* Patients with nontoxic/subtoxic nodular goiter confirmed by ultrasonography
* Patients with toxic nodular goiter
* Patients with Graves' disease

Exclusion Criteria:

* Treatment with drugs that alter thyroid function or size (the last 3 months prior to inclusion)
* Prior 131I treatment
* Alcohol, medicine or drug abuse
* Pregnancy or lactation
* No safe contraception
* Participation in another clinical trial
* Allergic reaction towards rhTSH
* Fine needle biopsy without valid diagnostic criteria for benign disease
* Suspicion of malignancy, increased ionized serum calcium and/or serum calcitonin
* Incontinence
* Physically or psychic condition that hinders corporation
* Ischemic attack up till 3 months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2002-04; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Ultrasonography/MR of the thyroid gland/benign goiter, in order to determine thyroid size after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Viveque Egsgaard Nielsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Result] Nielsen VE, Bonnema SJ, Boel-Jorgensen H, Grupe P, Hegedus L. Stimulation with 0.3-mg recombinant human thyrotropin prior to iodine 131 therapy to improve the size reduction of benign nontoxic nodular goiter: a prospective randomized double-blind trial. Arch Intern Med. 2006 Jul 24;166(14):1476-82. doi: 10.1001/archinte.166.14.1476. PMID 16864757